CLINICAL TRIAL: NCT05923567
Title: Novel Predictive Strategy Using CA19-9 and Fecal Elastase Levels to Make Treatment Decisions for Resectable Pancreatic Cancer; Retrospective Study
Brief Title: New Predictive Marker for Pancreatic Cancer Using CA19-9 and Fecal Elastase
Status: Active, not recruiting | Type: Observational
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Hyung Sun Kim, Assoiciate Professor, Gangnam Severance Hospital
Other Study IDs: 3-2020-0522
Record Dates: First submitted 2023-06-16; First posted 2023-06-28 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Paancreatic Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- CA19-9<385 & FE-1>100
- CA19-9<385 and FE-1>100
- CA19-9>385 & FE-1>100
- CA19-9>385 & FE-1<100

SUMMARY:
Background Carbohydrate antigen 19-9 (CA19-9) is used as a marker to predict recurrence and survival of patients with Pancreatic cancer(PDAC). Recently, fecal elastase-1(FE-1), a marker of pancreatic exocrine function, has been shown to correlate with prognosis in patients with PDAC. However, there have been no studies that have predicted prognosis by combining these two factors. In this study, investigators developed a predictive strategy for prognosis of PDAC using data on preoperative CA19-9 and FE-1 levels.6

Methods The clinical data of patients with resectable pancreatic cancer from two hospitals were analyzed. The cut-off points of preoperative CA19-9 and FE-1 levels were extracted from the Youden index and previous studies (385 U/ml and 100 µg/g stool, respectively). Cox proportional hazard models were used to investigate the association between preoperative tumor marker levels and survival (3-overall survival and 1-year recurrence free survival) after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Investigators conducted a retrospective study using data from 857 patients with pancreatic cancer enrolled in two hospitals in the Republic of Korea (179 from Gangnam Severance Hospital and 678 from Seoul National University Hospital) from January 5, 2010 to December 31, 2019.

Exclusion Criteria:

* Investigators excluded patients without information about preoperative tumor marker levels (n = 45), those who received neoadjuvant (n = 169), those with preoperative CA19-9 levels < 9.0 [Lewis antibody-negative patients] (n = 98), those with missing covariates (n = 3) and R2 resection (n = 6).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The clinical data of patients with resectable pancreatic cancer from two hospitals were analyzed. The cut-off points of preoperative CA19-9 and FE-1 levels were extracted from the Youden index and previous studies (385 U/ml and 100 µg/g stool, respectively). Cox proportional hazard models were used to investigate the association between preoperative tumor marker levels and survival (3-overall survival and 1-year recurrence free survival) after surgery.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-02-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
3yr overall survival | Survival period from surgery date, 3 years
  3-year survival rate for patients who underwent surgery for pancreatic cancer

SECONDARY OUTCOMES:
1yr disease free survival | Period without recurrence from the date of surgery, one year
  Recurrence rate in patients who have undergone surgery for pancreatic cancer within a year

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea